CLINICAL TRIAL: NCT00233909
Title: An Open-Label, Phase I/II Trial of Gemtuzumab Ozogamicin (GO) in Combination With Zosuquidar in Patients With CD33 Positive Acute Myeloid Leukemia
Brief Title: A Trial of Gemtuzumab Ozogamicin (GO) in Combination With Zosuquidar in Patients With CD33 Positive Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kanisa Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAN-979-02
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Leukemia, Myeloid
Keywords: Leukemia, Myeloid; Relapse; Chemotherapy; Zosuquidar; gemtuzumab ozogamicin (GO)
MeSH Terms: conditions — Leukemia, Myeloid; Recurrence | interventions — zosuquidar trihydrochloride; Gemtuzumab

INTERVENTIONS:
Drug: Zosuquidar
Drug: gemtuzumab ozogamicin

SUMMARY:
Chemotherapy drugs use different ways to stop cancer cells from dividing so they stop growing or die. Zosuquidar may help Gemtuzumab Ozogamicin (GO) kill more cancer cells by making cancer cells more sensitive to the drug. It is not known whether Gemtuzumab Ozogamicin (GO) is more effective with or without zosuquidar in treating acute myeloid leukemia.

DETAILED DESCRIPTION:
Purpose:

Phase I: Determine the optimal dose and schedule of GO and zosuquidar when used in combination.

Phase II: Determine the complete remission rate (CR+CRp)

ELIGIBILITY:
Inclusion Criteria:

1. Morphologic evidence of acute myeloid leukemia in first relapse.
2. Phase I: 18 years or older, Phase II: 50 years or older

Exclusion Criteria:

1. Prior treatment with zosuquidar
2. Any investigational agent within 1 month of enrollment and lack of recovery from toxicities secondary to those agents
3. History of stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

REFERENCES:
- [Derived] Marcelletti JF, Sikic BI. A clinical trial of zosuquidar plus gemtuzumab ozogamicin (GO) in relapsed or refractory acute myeloid leukemia (RR AML): evidence of efficacy based on leukemic blast P-glycoprotein functional phenotype. Cancer Chemother Pharmacol. 2023 Nov;92(5):369-380. doi: 10.1007/s00280-023-04578-9. Epub 2023 Aug 21. PMID 37603048